CLINICAL TRIAL: NCT07218393
Title: Retrospective and Prospective Real-World Evidence (RWE) Study Investigating Diagnosis and Therapeutic Management of Patients With HAE Type I or II in the Current Medical Practice in Egypt: the EXPLORHAE Study (EXPLORing Prospective and Retrospective Health Assessments of HAE in Egypt)
Brief Title: A Study About the Diagnosis and Management of Hereditary Angioedema (HAE) in Egypt
Acronym: EXPLORHAE
Status: Not yet recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-743-4031
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Phase: All participants who were diagnosed with HAE-C1INH type1 or type2 from January 2015 to August 2025; retrospective clinical data will be extracted for 5 months exclusively from patients' medical charts, and no direct patient interaction will occur.
  Interventions: Other: No intervention
- Prospective Phase: All participants with any newly diagnosed or admitted or follow-up HAE-C1INH type1 or type2; prospective clinical data will be actively collected over 12 months through routine visits and electronic data capture (EDC) entries.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a non-interventional study.

SUMMARY:
Hereditary angioedema (HAE) is a rare condition. It causes sudden swelling under the skin and inside the body, like in the belly, throat, or genitals. This swelling happens because of a temporary leak in blood vessels. HAE is classified based on the amount of a protein in the blood called C1 inhibitor (C1-INH): HAE with normal C1-INH levels and HAE with limited or insufficient C1-INH levels (C1-INH deficiency); HAE with C1-INH deficiency can be divided into Type1, with low levels of C1-INH, and Type 2, in which the protein is there, but does not work properly. This study will look at people with HAE Type1 or Type2.

The main aim of this study is to describe the diagnosis and management of people with HAE Type1 or HAE Type2 in Egypt. Other aims are to learn more about people with HAE Type1 or Type2, including, but not limited to, other conditions they may have, family history, impact of HAE on daily life, if treatment is stopped and the reasons.

During the study, information from already existing data in a participant's medical record will be reviewed and new data will be collected during routine visits of a participant to the study clinic.

ELIGIBILITY:
Inclusion Criteria: Retrospective Phase:

1. The participant has a confirmed HAE-C1INH type1 or type2 diagnosis in medical records (based on clinical history and/or laboratory diagnosis in medical records).
2. The participant was diagnosed and/or treated from January 2015 to August 2025.

Inclusion Criteria: Prospective Phase:

1. The participant has a physician-confirmed HAE-C1INH type1 or type2 diagnosis (based on clinical history and/or laboratory diagnosis).
2. The participant signed an informed consent or assent.
3. The participant should have had at least one visit to the treating physician/investigator during enrollment and the follow-up period.
4. The participant was not enrolled in the study's retrospective phase.

Exclusion Criteria: (For both retrospective and prospective phases):

1. Participant with AAE-C1INH (acquired angioedema), drug-induced angioedema (AE-DI) (example angiotensin-converting enzyme inhibitors-I [ACE-I] angioedema), allergic mediated angioedema, inflammatory angioedema, or idiopathic angioedema.
2. HAE participants with normal C1-INH (HAE-nC1INH).
3. Participant deemed unsuitable for participation for any reason, based on the investigator's clinical judgment.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric participants with HAE-C1INH type1 or type2, treated within a routine clinical setting in Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Age of Participants at Diagnosis (in years) of HAE-C1INH Type1 or Type2 | At Day 1
Percentage of Participants With HAE-C1INH Type1 or Type2 | At Day 1
Number and Type of First Symptom at Initial Manifestation | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With First Symptom at Initial Manifestation | Up to 5 months retrospectively, up to 12 months prospectively
Duration of First Symptom at Initial Manifestation | Up to 5 months retrospectively, up to 12 months prospectively
Number and Type of Confirmed Diagnosis of HAE-C1INH Type1 or Type2 | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Confirmed Diagnosis of HAE-C1INH Type1 or Type2 | Up to 5 months retrospectively, up to 12 months prospectively
Duration of Confirmed Diagnosis of HAE-C1INH Type1 or Type2 | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants with Recorded Diagnostic Test Results for C1-INH Antigenic Level, Serum Complement Component 4 (C4) Level, and C1-INH Functional Level | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants Receiving On-demand (OD), Short-term prophylaxis (STP), and Multiple Long-Term Prophylaxis (LTP) Therapies | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants who Received Prescriptions for Therapeutic Management With HAE-C1INH Type1 or Type2 | Up to 5 months retrospectively, up to 12 months prospectively
Number of Treatment Options Used for the Therapeutic Management of Participants With HAE-C1INH Type1 or Type2 | Up to 5 months retrospectively, up to 12 months prospectively
Number of Routes of Administration Used for the Therapeutic Management of Participants With HAE-C1INH Type1 or Type2 | Up to 5 months retrospectively, up to 12 months prospectively
Number of Dose Regimens Used for the Therapeutic Management of Participants With HAE-C1INH Type1 or Type2 | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants Switching Treatment for the Therapeutic Management of Participants With HAE-C1INH Type1 or Type2 | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Frequency of Treatment Changes for the Therapeutic Management of Participants With HAE-C1INH Type1 or Type2 | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Reason for Switching Treatment for the Therapeutic Management of Participants With HAE-C1INH Type1 or Type2 | Up to 5 months retrospectively, up to 12 months prospectively

SECONDARY OUTCOMES:
Number of Participants With Clinical Symptoms of HAE-C1INH Type1 or Type2 at Last Clinical Appointment | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Clinical Symptom Types of HAE-C1INH Type1 or Type2 at Last Clinical Appointment | Up to 5 months retrospectively, up to 12 months prospectively
Duration of Clinical Symptoms of HAE-C1INH Type1 or Type2 at Last Clinical Appointment | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Known Triggers at Diagnosis | Up to 5 months retrospectively, up to 12 months prospectively
  Triggers include stress, trauma, infection, contraception, menstruation, medication, food, burns, surgical procedures, and others.
Number of Participants With History of Upper Airway Edema | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With History of Abdominal Surgery due to HAE Misdiagnosis | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With HAE-related Death | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Response to Standard Allergy Medications | Up to 5 months retrospectively, up to 12 months prospectively
  Standard allergy medications (e.g. antihistamines, glucocorticoids, and epinephrine) that will be reported based on the symptom improvement, time to relief, reduction in symptom severity, and need for additional interventions.
Number of Participants With Presence of Comorbidities | Up to 5 months retrospectively, up to 12 months prospectively
Average Number of HAE Attacks per Month | Up to 5 months retrospectively, up to 12 months prospectively
Average Number of Attacks Requiring Acute Treatment per Month | Up to 5 months retrospectively, up to 12 months prospectively
Average Number of Attacks Requiring Emergency Care or Hospitalization per Month | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Severity of HAE Attack per Each Attack | Up to 5 months retrospectively, up to 12 months prospectively
  Number of participants with severity of HAE attack (mild, moderate, severe as reported or documented) per each attack.
Time of HAE Attack(s) at Each Onset During Follow-Up Visits or Date of Last Recorded HAE Attack | Up to 5 months retrospectively, up to 12 months prospectively
Duration of Symptoms for Each HAE Attack Onset During Subsequent Follow-Up Visits | Up to 5 months retrospectively, up to 12 months prospectively
Number of HAE Attacks per Month | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants Categorized by HAE Attack Characteristics | Up to 5 months retrospectively, up to 12 months prospectively
  HAE attack characteristics will include most common attack site(s) (e.g., abdominal, cutaneous, laryngeal), number of recurrent abdominal attacks, site of attack per each attack onset for each subsequent follow-up visit, and symptoms experienced per attack (e.g., pain, swelling, nausea).
Number of Participants With Prodromal Symptom | Up to 5 months retrospectively, up to 12 months prospectively
  Prodromal symptoms before attacks such as general discomfort, tiredness, irritability, skin symptoms, rash, and paresthesia per each attack onset for each subsequent follow-up visit will be reported.
Number of Participants With any Known Triggers Identified by the Participant as Related to the Onset of the Attack per Each Attack Onset for Each Subsequent Follow-up Visits | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With On-demand Treatment Medication for Each HAE Attack | Up to 5 months retrospectively, up to 12 months prospectively
Number and Type of Hospitalizations due to HAE Attacks | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Life-threatening Attacks | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants (Family Members) Diagnosed With HAE-C1INH Type1 or Type2 | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Degree of Relation (Parent, Sibling, Child) to Diagnosed Family Members | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Presence of Laryngeal or Life-threatening Attacks in Relatives | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Rate of Testing and of Diagnosis Among Tested Family Members | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With History of HAE-related Deaths in the Family | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participant's Relatives who Underwent Clinical and/or Lab Assessment for HAE diagnosis | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Clinical Assessment for HAE Diagnosis With Symptoms Description for the Patient, their Descendants, or Relatives | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Laboratory Testing for the Participant, Their Descendants, or Relatives | Up to 5 months retrospectively, up to 12 months prospectively
Number of Follow-up Visits Routinely Performed (Average per Year) During the Retrospective and Prospective Phase | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants Who Missed Days at Work or School and Social Life due to HAE Attack | Up to 5 months retrospectively, up to 12 months prospectively
Number of Participants With Treatment Discontinuation | Up to 5 months retrospectively, up to 12 months prospectively
  Participants who discontinued the treatment due to reasons such as lack of efficacy, safety concerns, compliance issues, or others.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (7):
- Egypt (7):
  - Mansoura university hospital, Al Mansurah
  - Alexandria university_Clinical Research Center, Alexandria
  - Ain shams university hospital_Pediatrics, Cairo
  - Ain shams university hospital, Cairo
  - Cairo university hospital_Pediatrics, Giza
  - Cairo university hospital, Giza
  - Zagazig university hospital, Zagazig

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/e36bb72fdb9e4ed8??page=1&idFilter=TAK-743-4031